CLINICAL TRIAL: NCT06109532
Title: Prevalence of Hyponatremia in Dengue Infected Patients: Relationship With Systemic Inflammation.
Acronym: HINDIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Nacional Profesor Alejandro Posadas (Other)
Responsible Party: Principal Investigator, Ladislao Diaz Ballve, Principal Investigator, Hospital Nacional Profesor Alejandro Posadas
Other Study IDs: HINDIP162023
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Hyponatremia; Dengue; Inflammation
Keywords: HYPONATREMIA; DENGUE; INFLAMMATION
MeSH Terms: conditions — Hyponatremia; Dengue; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DENGUE INFECTED PATIENTS. YEAR 2016: We conducted a prospective cohort study in patients with newly diagnosed dengue infection at Hospital Posadas in Argentina, between January 1, 2016, and december 31, 2016. Diagnosis was confirmed by IgM serology or PCR. Hyponatremia was defined as serum sodium concentration ≤135 mEq/L.
  Interventions: Other: hyponatremia
- DENGUE INFECTED PATIENTS. YEAR 2020: We conducted a prospective cohort study in patients with newly diagnosed dengue infection at Hospital Posadas in Argentina, between January 1, 2020, and december 31, 2020. Diagnosis was confirmed by IgM serology or PCR. Hyponatremia was defined as serum sodium concentration ≤135 mEq/L.
  Interventions: Other: hyponatremia
- DENGUE INFECTED PATIENTS. YEAR 2023: We conducted a prospective cohort study in patients with newly diagnosed dengue infection at Hospital Posadas in Argentina, between January 1, 2023, and november 1, 2023. Diagnosis was confirmed by IgM serology or PCR. Hyponatremia was defined as serum sodium concentration ≤135 mEq/L.
  Interventions: Other: hyponatremia

INTERVENTIONS:
Other: hyponatremia — hyponatremia at admission in dengue infected patients

SUMMARY:
Prospective cohort study in patients with newly diagnosed dengue infection at Hospital Posadas in Argentina, between January 1, 2016, and November 1, 2023. Diagnosis was confirmed by IgM serology or PCR. Hyponatremia was defined as serum sodium concentration ≤135 mEq/L.

DETAILED DESCRIPTION:
Background Dengue infection is becoming more prevalent worldwide and is associated with systemic inflammation. Systemic Inflammation is associated with non-osmotic release of ADH.

Methods: Participants conducted a prospective cohort study in patients with newly diagnosed dengue infection at Hospital Posadas in Argentina, between January 1, 2016, and November 1, 2023. Diagnosis was confirmed by IgM serology or PCR. Hyponatremia was defined as serum sodium concentration ≤135 mEq/L.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis confirmed by PCR, non structural protein 1 (NS1) antigen or IgM serology.

Plasma sodium at admission.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed dengue infection at Hospital Posadas in Argentina, between January 1, 2016, and May 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Admission to the hospital | between january 1, 2023 and november 1, 2023
  Risk for admission to the hospital

CONTACTS AND LOCATIONS:
Overall Officials: CARLOS EGHI, MD, Principal Investigator — HOSPITAL NACIONAL PROF. A. POSADAS
Locations (2):
- Argentina (2):
  - Ladislao Diaz Ballve, Haedo, Buenos Aires
  - Hospital Posadas, Buenos Aires

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ayus JC, Negri AL, Moritz ML, Lee KM, Caputo D, Borda ME, Go AS, Eghi C. Hyponatremia, Inflammation at Admission, and Mortality in Hospitalized COVID-19 Patients: A Prospective Cohort Study. Front Med (Lausanne). 2021 Dec 2;8:748364. doi: 10.3389/fmed.2021.748364. eCollection 2021. PMID 34926496